CLINICAL TRIAL: NCT07155681
Title: Evaluating Healthcare Professionals' Satisfaction and Stress Mitigation Using Virtual Reality Intervention in Surgical Ward: a Multination Feasibility Study
Brief Title: Evaluating Healthcare Professionals' Satisfaction and Stress Mitigation Using Virtual Reality Intervention in Surgical Ward
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: European Union (Horizon Europe Programme) (Unknown); Rigshospitalet, Denmark (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Sophie Vermeulen, Medical doctor, PhD Candidate Department of Surgery, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025.0425
Record Dates: First submitted 2025-08-17; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Stress; Stress (Psychology)
Keywords: VR; Virtual Reality; Stress; Resilience; Healthcare professionals; healthcare workers; nurses; hospital; surgical ward

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR intervention (Experimental)
  Interventions: Device: Virtual Reality intervention

INTERVENTIONS:
Device: Virtual Reality intervention — Virtual Realtiy intervention with biofeedback for 10 minutes during a shift on the ward for healthcare professionals

SUMMARY:
The goal of this feasibility study is to learn whether a VR intervention is feasible, acceptable, and satisfactory for healthcare workers in surgical wards to help mitigate stress. Secondary objectives include assessing its potential contribution to stress reduction, user comfort, and practical integration into daily workflows.

Participants will take part in a single 10-minute VR intervention session.

DETAILED DESCRIPTION:
This study investigates the use of the HealthyMind Virtual Reality (VR) application as an innovative intervention to reduce stress among healthcare workers in surgical departments. Although workplace stress is common, there is currently a lack of structured interventions to address it.

The VR application provides healthcare professionals with the opportunity to relax through immersive, calming three-dimensional environments, such as a sunset by the sea or a mountain landscape. The VR headset is paired with an armband that non-invasively measures physiological parameters, including heart rate and heart rate variability. Based on these data, the VR environment automatically adapts to the user's stress level, for example by introducing a guided breathing exercise.

The intervention can be used at any self-selected moment during a shift, with the aim of offering a short and effective recovery break. The primary aim of this study is to evaluate the feasibility, acceptability, and user satisfaction of the VR intervention among healthcare workers. Secondary objectives include assessing its potential contribution to stress reduction, user comfort, and practical integration into daily workflows.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering healthcare professionals (≥18 years old) working in direct patient care, such as nurses, residents, physician assistants, and surgeons, on the surgical ward.

Exclusion Criteria:

* Diagnosed with epilepsy
* Experienced VR as a trigger for their migraines
* Severe dizziness, nausea or physical disabilities will be excluded.
* Diagnosed with arrythmias, bradycardia or tachycardia
* Not able to wear the VR headset due to physical or psychological conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
AIM-IAM-FIM • Acceptability of Intervention Measure (AIM), • Intervention Appropriateness Measure (IAM), • Feasibility of Intervention Measure (FIM) | Immediately after the VR intervention the scale will be filled in by the participant
  Each subscale comprises four elements ranging from 1 (completely disagree) to 5 (completely agree)
User satisfaction | Immediately after the VR intervention
  NRS score ranging from 0 (not satisfied) to 10 (very satisfied)

SECONDARY OUTCOMES:
Stress level | immediately before the intervention (pre-intervention) and immediately after the intervention (post-intervention)
  NRS score ranging from 0 (not satisfied) to 10 (very satisfied)
CSQ-VR | immediately after the VR intervention
  Assessing user comfort with the CyberSickness in Virtual Reality Questionnaire (CSQ-VR). With a likert scale ranging from 1 = absent feeling to 7 = extreme feeling. with higher scores indicating more discomfort
Best organizational fit | At a scheduled moment within 1 month after the intervention
  Using a qualitative semi-structured follow-up interview after completing the experience in five participants per center.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Eskes, associate professor, Principal Investigator — AmsterdamUMC
Locations (2):
- Rhigshospitalet, Copenhagen, Denmark
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: a link to the KEEPCARING website. This study is part of the project — https://keepcaring.eu